CLINICAL TRIAL: NCT04920708
Title: Randomised Phase II Study of Induction Fulvestrant and CDK4/6 Inhibition With the Addition of Ipatasertib in Metastatic ER+/HER2- Breast Cancer Patients Without ctDNA Suppression
Brief Title: Fulvestrant, Ipatasertib and CDK4/6 Inhibition in Metastatic ER+/HER2- Breast Cancer Patients Without ctDNA Suppression
Acronym: FAIM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Pfizer (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR5214
Record Dates: First submitted 2021-05-27; First posted 2021-06-10 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Breast Cancer; ER+ Breast Cancer; Advanced Breast Cancer
Keywords: Fulvestrant; Palbociclib; Ipatasertib; ctDNA
MeSH Terms: conditions — Breast Neoplasms | interventions — ipatasertib; Fulvestrant; palbociclib; abemaciclib; ribociclib

STUDY DESIGN:
Intervention Model Description: Patients starting standard of care CDK4/6 inhibitors and fulvestrant will have ctDNA assessment at Cycle 1 Day 1 (C1D1) and Cycle 1 Day 15 (C1D15).
  Patients with high ctDNA levels at C1D15 will be randomised in a 1:1 ratio to palbociclib + fulvestrant (comparison arm) or palbociclib + fulvestrant + ipatasertib (interventional arm).
  Patients with ctDNA suppressed at C1D15 will continue standard of care, fulvestrant+CDK4/6 inhibitor (observational arm). The first 100 patients of this group will be followed for PFS, OS and ctDNA collection.
  Patients with no detectable ctDNA at screening will continue on standard of care. The first 50 of this group will be followed for PFS, OS, time to next treatment, and time to chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Palbociclib + Fulvestrant + Ipatasertib (Interventional arm) (Experimental): Where high ctDNA is detected in screening, patients to be randomised on a 1:1 basis to interventional arm or comparison arm. Patients randomised to interventional arm receive Palbociclib + Fulvestrant + Ipatasertib. n = 87.
  Interventions: Drug: Ipatasertib 300mg; Drug: Fulvestrant 500g; Drug: Palbociclib 75mg-125mg
- Palbociclib + Fulvestrant (Comparison arm) (Active Comparator): Where high ctDNA is detected in screening, patients to be randomised on a 1:1 basis to interventional arm or comparison arm. Patients randomised to Comparison arm receive Palbociclib + Fulvestrant. n = 87.
  Interventions: Drug: Fulvestrant 500g; Drug: Palbociclib 75mg-125mg
- Standard of Care (No ctDNA observational arm) (Active Comparator): Where no ctDNA is detected in screening, patients to be allocated to the observational arm and receive standard of care (Abemaciclib / Ribociclib / Palbociclib + fulvestrant). n = 50.
  Interventions: Drug: Fulvestrant 500g; Drug: CDK4/6 Inhibitor
- Standard of Care (Low ctDNA observational arm) (Active Comparator): Where low ctDNA is detected in screening, patients to be allocated to the observational arm and receive standard of care (Abemaciclib / Ribociclib / Palbociclib + fulvestrant). n = 100.
  Interventions: Drug: Fulvestrant 500g; Drug: CDK4/6 Inhibitor

INTERVENTIONS:
Drug: Ipatasertib 300mg — Ipatasertib 300mg once daily. Oral administration. Treatment is continuous daily for 21 days, followed by 7 days off, to complete a 28 day cycle.
  Other Names: RG7440
  Arms: Palbociclib + Fulvestrant + Ipatasertib (Interventional arm)
Drug: Fulvestrant 500g — Fulvestrant 500mg administered intramuscularly in the buttocks slowly (1-2 minutes per injection) as two 5-mL injections (one in each buttock). Administered days 1 and 15 of Cycle 1. For subsequent cycles, patients will receive fulvestrant as described above in the clinic on Day 1 of each cycle or approximately every 4 weeks.
  Other Names: Faslodex
Drug: Palbociclib 75mg-125mg — Palboclicib 75mg-125mg once daily, dependent on toxicities. Oral administration. Treatment is continuous daily for 21 days, followed by 7 days off, to complete a 28 day cycle.
  Other Names: Ibrance
  Arms: Palbociclib + Fulvestrant (Comparison arm); Palbociclib + Fulvestrant + Ipatasertib (Interventional arm)
Drug: CDK4/6 Inhibitor — CDK4/6 inhibitor. As per current standard of care regime for ER+/HER2- breast cancer.
  Other Names: Abemaciclib / Ribociclib / Palbociclib
  Arms: Standard of Care (Low ctDNA observational arm); Standard of Care (No ctDNA observational arm)

SUMMARY:
Analysis of circulating tumour DNA (ctDNA) found in a patient's peripheral blood can identify cancer progression and predict a patient's response to therapy. By using ctDNA analysis and imaging techniques, the FAIM trial aims to determine whether the addition of the experimental drug ipatasertib to a standard combination of the hormone treatment fulvestrant and the targeted agent palbociclib increases progression free survival (PFS) for patients with hormone-receptor positive and human epidermal growth factor receptor 2 negative (HR+/HER2-) breast cancer.

DETAILED DESCRIPTION:
Circulating tumour DNA (ctDNA) can be found in the peripheral blood of patients with cancer. ctDNA analysis provides a readily available, serial source of tumour DNA which can be used to monitor disease and predict a patients response to therapy.

Relative changes in ctDNA after 15 days of treatment with palbociclib and fulvestrant has been found to strongly predict progression free survival (PFS) in hormone-receptor positive and human epidermal growth factor receptor 2 negative (HR+/HER2-) breast cancer patients: patients without ctDNA suppression after 2 weeks of treatment had a significantly shorter PFS compared to those with ctDNA suppression, identifying a group of patients who require additional therapy to prevent early progression.

The FAIM trial is a randomised, open-label study which will aim to determine whether the addition of ipatasertib to standard of care CDK4/6 inhibitors + fulvestrant increases PFS in patients who lack ctDNA suppression after 15 days of treatment. Patients starting standard of care CDK4/6 inhibitors + fulvestrant will have a ctDNA assessment on cycle 1 day 1 (C1D1) and cycle 1 day 15 (C1D15). Those with high ctDNA levels at C1D15 will be randomised on a 1:1 basis to either standard of care (CDK4/6 inhibitors + fulvestrant) or standard of care plus the experimental drug ipatasertib (CDK4/6 inhibitor + fulvestrant + ipatasertib). Patients with ctDNA suppression at C1D15 will continue standard of care (fulvestrant+CDK4/6 inhibitor); the first 100 patients of this group will be followed for PFS and ctDNA collection. Patients without detectable ctDNA on C1D1 will be followed and treated according standard of care; the first 50 patients of this group will be followed for PFS, overall survival (OS), time to next treatment, and time to chemotherapy. Progression free survival will be monitored using RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of metastatic or inoperable locally advanced ER positive/HER2 negative breast cancer. Assessment of ER and HER2 status as per local assessment. Histologically proven primary ER+ (Allred score 3/8 or greater, or stain in >1% of cancer cells) and HER2- (immunohistochemistry 0/1+ or negative by in situ hybridization) breast cancer as determined by local laboratory.
2. Be willing to consent for an archival tumour tissue sample (of advanced disease) to be requested for transfer to the Royal Marsden for future review during study screening. Patients without a metastatic biopsy may be eligible if archival tumour from the breast primary tumour is available, but only after discussion with the Chief Investigator.
3. Previously treated with no more than one prior line of chemotherapy for advanced disease.
4. Patients eligible according to standard of care for fulvestrant in combination with a CDK4/6 inhibitor (abemaciclib, palbociclib, or ribociclib).
5. Patients must have received at least one prior line of hormone therapy for advanced disease and progressed on or within 1 month from stopping prior endocrine therapy for advanced disease, or relapsed on or within 12 months of completing adjuvant endocrine therapy.
6. Measurable disease (RECIST 1.1) or assessable bone disease (lytic or mixed lytic sclerotic).
7. Eastern Cooperative Oncology Group (ECOG) performance status 0,1 or 2.
8. Estimated life expectancy of at least 3 months.
9. Adequate bone marrow, renal, and liver function within 14 days before the first study treatment on Day 1 of Cycle 1, defined by the following:

   1. Neutrophils (ANC ≥ 1500/μL), Haemoglobin ≥9 g/dL, Platelet count ≥100,000/μL
   2. Serum albumin ≥3 g/dL
   3. Total bilirubin ≤1.5 x the upper limit of normal (ULN), with the following exception: patients with known Gilbert syndrome who have serum bilirubin ≤3 x ULN may be enrolled
   4. AST and ALT ≤2.5 x ULN, with the following exception: patients with documented liver or bone metastases may have AST and ALT ≤5 x ULN.
   5. ALP ≤2 x ULN, with the following exceptions: patients with known liver involvement may have ALP ≤5 x ULN, patients with known bone involvement may have ALP ≤7 x ULN
   6. Serum creatinine ≤1.5 x ULN or creatinine clearance ≥50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation.
   7. INR <1.5 x ULN and aPTT <1.5 x ULN. Patients requiring formal anticoagulation should receive either low-molecular weight heparin or a direct oral anticoagulant.
10. Fasting glucose ≤150mg/dL and HbA1c ≤7.5%.
11. Negative serum pregnancy test at screening (females of childbearing potential).
12. Patients able to have children must agree to use two highly effective methods of contraception throughout the study and for 2 years after last dose of fulvestrant and at least two years after last dose. Patients must additionally agree to refrain from donating eggs during this period.
13. Signed and dated informed consent.
14. Patients willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other procedures.
15. Pre/peri-menopausal patients must be treated with GnRH agonist beginning at least 7 days prior to Day 1 of Cycle 1 and continuing every 28 days for the duration of study treatment.

Exclusion Criteria:

1. Previous fulvestrant and/or CDK4/6 inhibitor (abemaciclib, palbociclib or ribociclib) in any setting.
2. Prior use of AKT inhibitor (any setting).
3. History of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills.
4. Systemic chemotherapy within 14 days prior to study entry.
5. Major surgery within 4 weeks or radiation therapy within 14 days prior to study entry.
6. Patients with known leptomeningeal disease, symptomatic brain metastases requiring steroids, untreated brain metastases or spinal cord compression.
7. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality including any of the following:

   1. History of angina pectoris, symptomatic pericarditis, coronary artery bypass graft (CABG) or myocardial infarction within 12 months prior to study entry.
   2. Known (documented) cardiomyopathy, i.e known left ventricular ejection fraction (LVEF) < 50% (ECHO or MUGA not needed specifically for this trial).
   3. History of symptomatic cardiac failure (NYHA class II-IV or LVEF <50%), uncontrolled hypertension, cardiac dysrhythmia including atrial fibrillation requiring medication, significant/symptomatic bradycardia, Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome or any of the following:, cerebrovascular accident, or transient ischemic attack within 12 months; known risk factors for prolonged QT interval or Torsade's de Pointes; Uncorrected hypomagnesaemia or hypokalaemia of Grade 3 or higher; Systolic Blood Pressure (SBP) >160 mmHg or <90 mmHg; Bradycardia (heart rate <50 at rest), by ECG (based on a mean of 3 ECGs) or pulse; On screening, QTcF >470 screening ECG (based on a mean of 3 ECGs).
8. Pneumonitis, interstitial lung disease or pulmonary fibrosis.
9. Type I or II diabetes requiring insulin.
10. Use of drugs that are known potent cytochrome P450 3A inducers or inhibitors within 2 weeks or 5 elimination half-lives (whichever is longer) before the first dose of study drug.
11. Known HIV or AIDS-related illness.
12. Active infection requiring systemic therapy.
13. Known positive HBV or HCV test indicating acute or chronic infection

    1. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible.
    2. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
14. Clinically significant liver disease consistent with Child Pugh class B or C.
15. Administration of a live vaccine within 4 weeks prior to study entry.
16. Diagnosis of other malignancy within 5 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or cervix.
17. Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry and/or during study participation.
18. Persisting toxicity related to prior therapy >Grade 1 (except for stable peripheral neuropathy grade 2 or alopecia grade 2).
19. Other severe acute or chronic medical condition, including colitis, inflammatory bowel disease, psychiatric condition, recent or active suicidal ideation or behaviour, or end stage renal disease on haemodialysis, or laboratory abnormality that may increase the risk associated with study participation or investigational products administration or may interfere with the interpretation of results and, in the judgment of the Investigator, would make the patient inappropriate study entry.
20. Radiation therapy (other than palliative radiation to bony metastases) as cancer therapy within 4 weeks prior to initiation of study treatment.
21. Palliative radiation to bony metastases within 2 weeks prior to initiation of study treatment.
22. Allergy or hypersensitivity to components of the ipatasertib, palbociclib, or fulvestrant.
23. Patients able to have children who are unwilling or unable to use 2 highly effective method(s)¹ of contraception for the duration of the study and for at least 60 days after the last dose of investigational product. Patient pregnant or breastfeeding.
24. Need for chronic corticosteroid therapy of >10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressants for a chronic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Assess progression free survival (PFS) | Time from date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 38 months
  To compare PFS in patients randomised between palbociclib/fulvestrant/ipatasertib versus standard of care palbociclib-fulvestrant alone, in advanced ER+/HER2- breast cancer patients with trackable mutations and high ctDNA after 2 weeks of CDK4/6 inhibitor/fulvestrant.

SECONDARY OUTCOMES:
Use NCI CTCAE V5.0 to assess safety and tolerability of palbociclib/fulvestrant/ipatasertib compared to palbociclib/fulvestrant alone | 36 months (treatment duration + follow-up duration)
  • To assess the overall safety and tolerability of palbociclib/fulvestrant/ipatasertib compared to standard of care palbociclib/fulvestrant alone. Safety will be evaluated continuously using NCI CTCAE V5.0.
Assess overall survival | 36 months (treatment duration + follow-up duration)
  • To assess overall survival in patients receiving palbociclib/fulvestrant/ipatasertib compared to standard of care palbociclib/fulvestrant alone
Assess objective response rate | 36 months (treatment duration + follow-up duration)
  • To assess the objective response rate in patients receiving palbociclib/fulvestrant/ipatasertib compared to standard of care palbociclib/fulvestrant alone
Report progression free survival (PFS) in patients with low ctDNA and high ctDNA | Time from date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 38 months
  • To report PFS in patients with high ctDNA randomised to standard of care palbociclib/fulvestrant alone with those with suppressed ctDNA on standard of care CDK4/6 inhibitor/fulvestrant alone (observational arm)
Compare progression free survival (PFS) in the subgroup of advanced ER+/HER2- breast cancer patients | Time from date of randomisation until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 38 months
  o compare PFS in patients randomised between palbociclib/fulvestrant/ipatasertib and palbociclib/fulvestrant alone, in the subgroup of advanced ER+/HER2- breast cancer patients with PIK3CA/PTEN/AKT1 mutations or PTEN loss and high ctDNA on palbociclib/fulvestrant

OTHER OUTCOMES:
Evaluate changes in ctDNA in patients with high ctDNA C1D15 | 36 months (treatment duration + follow-up duration)
  • To evaluate changes in ctDNA in patients randomised to palbociclib/fulvestrant/ipatasertib or standard of care palbociclib/fulvestrant alone.
Compare progression free survival (PFS) in patients with high ctDNA at C1D15 and genetic alterations identified in ctDNA sequencing. | 36 months (treatment duration + follow-up duration)
  • To compare PFS in patients randomised between SOC palbociclib/fulvestrant + /ipatasertib and SOC palbociclib/fulvestrant alone, in subgroups of advanced ER+/HER2- breast cancer patients with genetic alterations identified in ctDNA sequencing data.
Report progression free survival (PFS) in patients with undetectable ctDNA and those with detected ctDNA at C1D1 with and without suppression at C1D15. | 36 months (treatment duration + follow-up duration)
  • To compare report PFS in patients with undetectable ctDNA at Cycle 1 Day 1 and those with detectable ctDNA with and without ctDNA suppression at Day 15.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Okines, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (18):
- United Kingdom (18):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Royal Cornwall Hospital, Truro, Cornwall
  - Mount Vernon Cancer Centre, London, Surrey
  - Velindre Cancer Centre, Cardiff, Wales
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey NHS Foundation Trust, Guildford
  - University Hospitals of Leicester NHS Trust, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - Royal Free Hospital, London
  - Guy's and St Thomas's NHS Foundation Trust, London
  - Royal Marsden NHS Foundation Trust, London
  - Imperial College University Hospitals NHS Trust, London
  - University College London Hospital, London
  - Maidstone Oncology Centre, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Southampton Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: No
The confidentiality of patients participating in this trial will be protected and each participant will be assigned a unique trial number at the point of registration which will be used to identify eCRFs and anything else sent to the sponsor or other third parties. No patient identifiable data will be shared outside of the participating site.

REFERENCES:
- [Background] Turner NC, Ro J, Andre F, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Huang Bartlett C, Zhang K, Giorgetti C, Randolph S, Koehler M, Cristofanilli M; PALOMA3 Study Group. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Jul 16;373(3):209-19. doi: 10.1056/NEJMoa1505270. Epub 2015 Jun 1. PMID 26030518
- [Background] Turner NC, Slamon DJ, Ro J, Bondarenko I, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Andre F, Puyana Theall K, Huang X, Giorgetti C, Huang Bartlett C, Cristofanilli M. Overall Survival with Palbociclib and Fulvestrant in Advanced Breast Cancer. N Engl J Med. 2018 Nov 15;379(20):1926-1936. doi: 10.1056/NEJMoa1810527. Epub 2018 Oct 20. PMID 30345905
- [Background] Cristofanilli M, Turner NC, Bondarenko I, Ro J, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Zhang K, Theall KP, Jiang Y, Bartlett CH, Koehler M, Slamon D. Fulvestrant plus palbociclib versus fulvestrant plus placebo for treatment of hormone-receptor-positive, HER2-negative metastatic breast cancer that progressed on previous endocrine therapy (PALOMA-3): final analysis of the multicentre, double-blind, phase 3 randomised controlled trial. Lancet Oncol. 2016 Apr;17(4):425-439. doi: 10.1016/S1470-2045(15)00613-0. Epub 2016 Mar 3. PMID 26947331
- [Background] O'Leary B, Hrebien S, Morden JP, Beaney M, Fribbens C, Huang X, Liu Y, Bartlett CH, Koehler M, Cristofanilli M, Garcia-Murillas I, Bliss JM, Turner NC. Early circulating tumor DNA dynamics and clonal selection with palbociclib and fulvestrant for breast cancer. Nat Commun. 2018 Mar 1;9(1):896. doi: 10.1038/s41467-018-03215-x. PMID 29497091
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Telli ML, Gradishar WJ, Ward JH. NCCN Guidelines Updates: Breast Cancer. J Natl Compr Canc Netw. 2019 May 1;17(5.5):552-555. doi: 10.6004/jnccn.2019.5006. PMID 31117035
- [Background] Cardoso F, Senkus E, Costa A, Papadopoulos E, Aapro M, Andre F, Harbeck N, Aguilar Lopez B, Barrios CH, Bergh J, Biganzoli L, Boers-Doets CB, Cardoso MJ, Carey LA, Cortes J, Curigliano G, Dieras V, El Saghir NS, Eniu A, Fallowfield L, Francis PA, Gelmon K, Johnston SRD, Kaufman B, Koppikar S, Krop IE, Mayer M, Nakigudde G, Offersen BV, Ohno S, Pagani O, Paluch-Shimon S, Penault-Llorca F, Prat A, Rugo HS, Sledge GW, Spence D, Thomssen C, Vorobiof DA, Xu B, Norton L, Winer EP. 4th ESO-ESMO International Consensus Guidelines for Advanced Breast Cancer (ABC 4)dagger. Ann Oncol. 2018 Aug 1;29(8):1634-1657. doi: 10.1093/annonc/mdy192. No abstract available. PMID 30032243
- [Background] Johnston SR. Enhancing the efficacy of hormonal agents with selected targeted agents. Clin Breast Cancer. 2009 Jun;9 Suppl 1:S28-36. doi: 10.3816/CBC.2009.s.003. PMID 19561004
- [Background] Musgrove EA, Sutherland RL. Biological determinants of endocrine resistance in breast cancer. Nat Rev Cancer. 2009 Sep;9(9):631-43. doi: 10.1038/nrc2713. PMID 19701242
- [Background] Zardavas D, Irrthum A, Swanton C, Piccart M. Clinical management of breast cancer heterogeneity. Nat Rev Clin Oncol. 2015 Jul;12(7):381-94. doi: 10.1038/nrclinonc.2015.73. Epub 2015 Apr 21. PMID 25895611
- [Background] Meyerson M, Harlow E. Identification of G1 kinase activity for cdk6, a novel cyclin D partner. Mol Cell Biol. 1994 Mar;14(3):2077-86. doi: 10.1128/mcb.14.3.2077-2086.1994. PMID 8114739
- [Background] Coudreuse D, Nurse P. Driving the cell cycle with a minimal CDK control network. Nature. 2010 Dec 23;468(7327):1074-9. doi: 10.1038/nature09543. PMID 21179163
- [Background] O'Leary B, Finn RS, Turner NC. Treating cancer with selective CDK4/6 inhibitors. Nat Rev Clin Oncol. 2016 Jul;13(7):417-30. doi: 10.1038/nrclinonc.2016.26. Epub 2016 Mar 31. PMID 27030077
- [Background] Sledge GW Jr, Toi M, Neven P, Sohn J, Inoue K, Pivot X, Burdaeva O, Okera M, Masuda N, Kaufman PA, Koh H, Grischke EM, Frenzel M, Lin Y, Barriga S, Smith IC, Bourayou N, Llombart-Cussac A. MONARCH 2: Abemaciclib in Combination With Fulvestrant in Women With HR+/HER2- Advanced Breast Cancer Who Had Progressed While Receiving Endocrine Therapy. J Clin Oncol. 2017 Sep 1;35(25):2875-2884. doi: 10.1200/JCO.2017.73.7585. Epub 2017 Jun 3. PMID 28580882